CLINICAL TRIAL: NCT04607187
Title: Ultrasound B Mode Imaging and Elastography During Administration of Xiaflex (Collagenase Clostridium Histolyticum) for Dupuytren's Contracture: A Pilot Study (The UBIEX-DC Study)
Brief Title: Ultrasound B Mode Imaging and Elastography
Acronym: UBIEX-DC
Status: Completed | Type: Observational
Sponsor: Theresa Bass-Goldman (Other)
Collaborators: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Theresa Bass-Goldman, Principal Investigator Paul J. DeMarco, MD, Arthritis & Rheumatism Associates, P.C.
Organization: Arthritis & Rheumatism Associates, P.C. (Other)
Other Study IDs: 351-CRBR
Record Dates: First submitted 2013-11-22; First posted 2020-10-29 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Dupuytren's Contractures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Normals, Dupuytren's subjects with and without treatment: Ultrasound analysis of patient receiving treatment for Dupuytren's

SUMMARY:
A Pilot Study on Ultrasound B mode Imaging and Elastography during administration of Xiaflex (collagenase clostridium histolyticum) for Dupuytren's contracture.

DETAILED DESCRIPTION:
Ultrasound analysis will be obtained on patient that receives Xiaflex as standard of care for Dupuytren's contracture

ELIGIBILITY:
Inclusion Criteria:

* Normal Hand or Hand Dupuytren's contracture

Exclusion Criteria:

* Previous treatment of Dupuytren's cord

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Three groups of people will take part in the research:
  5-Normal subjects without a Dupuytren's contracture 5-Subjects that have a hand Dupuytren's contracture that will not receive tx 10-Subjects that have a hand Dupuytren's contracture that will receive tx
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Ultrasound B mode Imaging and Elastography | 30 day trial
  A Pilot Study: Ultrasound B mode Imaging and Elastography during administration of Xiaflex

CONTACTS AND LOCATIONS:
Locations (1):
- The Center for Rheumatology and Bone Research a division of Arthritis and Rheumatism Associates, P.C., Wheaton, Maryland, United States